CLINICAL TRIAL: NCT01229007
Title: A Phase III, Open-Label, Multicentre Study to Evaluate Efficacy, Pharmacokinetics, and Safety of Biostate® in Paediatric Subjects With Haemophilia A
Brief Title: Study of Biostate® in Children With Hemophilia A
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CSL Behring (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSLCT-BIO-08-53; 2009-015112-18 (EudraCT Number); 1495 (Other: CSL Behring)
Record Dates: First submitted 2010-10-01; First posted 2010-10-27 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2014-07

CONDITIONS: Hemophilia A
Keywords: Hemophilia A; Children
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Biostate (Experimental)
  Interventions: Biological: Biostate

INTERVENTIONS:
Biological: Biostate — 1 dose of 50 IU FVIII/kg body weight of Biostate administered intravenously on Day 1 in the PK component, followed by the Efficacy component for continuation of Biostate therapy, as required for a minimum of 50 exposure days.

SUMMARY:
The objective of this study is to assess the efficacy and safety of a Von Willebrand Factor/Factor VIII (VWF/FVIII), Biostate, and to investigate the pharmacokinetics of Biostate in children with haemophilia A.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects between 0 and <12 years of age.
* Diagnosed with severe haemophilia A (FVIII:C <1%), and pre-treated for a minimum of 20 to 50 exposure days.
* Have evidence of vaccination against hepatitis A and B (or presence of antibodies against hepatitis A and B due to either a previous infection or prior immunisation), as documented in the medical notes at enrolment.
* The subject and/or legal guardian understand(s) the nature of the study and has/have given written informed consent to participate in the study and is/are willing to comply with the protocol.

Exclusion Criteria:

* For all subjects at Day 1: Are actively bleeding.
* Have received an infusion of any FVIII product, cryoprecipitate, whole blood, plasma or desmopressin acetate in the 4 days prior to their dosing within the PK component.
* Have a known history of, or who are suspected of having FVIII inhibitors.
* Have received aspirin or other non-steroidal anti-inflammatory drugs (NSAIDs) within 7 days of administration of the IMP.
* Have an impaired liver function ie, bilirubin >1.5 x upper limit of normal (ULN) and/or aspartate/alanine aminotransferase (AST/ALT) >2.5 x ULN (referring to limits of the laboratory that performs the determination) at Screening.
* Are human immunodeficiency virus [HIV]-1/-2 antibody positive with a viral load of >200/µL.
* Suffer from an acute or chronic medical condition, other than haemophilia A, which may, in the opinion of the Investigator, affect the conduct of the study.
* Suffering from von Willebrand disease (VWD) with von Willebrand factor: ristocetin cofactor (VWF:RCo) level <50 IU/dL at Screening.
* Have a known or suspected hypersensitivity or previous evidence of severe side effects to a plasma-derived FVIII product or to human albumin.
* Have participated in a clinical study or used an investigational compound in another study (eg, a new chemical entity not registered for clinical use) in the 3 months preceding the first day of IMP administration, or are planning to enter such a study during the study period.
* Unwillingness and/or inability to comply with the study requirements.

Max Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2010-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Subjective assessment of Haemostatic efficacy | Over minimum of 50 exposure days
Incremental recovery of FVIII | Samples taken prior and then 0.5, 4, 8, 24, and 48 h after the infusion on Day 1
Half-life of FVIII | Samples taken prior and then 0.5, 4, 8, 24, and 48 h after the infusion on Day 1
Area under the concentration curve (AUC) of FVIII | Samples taken prior and then 0.5, 4, 8, 24, and 48 h after the infusion on Day 1
Mean residence time (MRT) of FVIII | Samples taken prior and then 0.5, 4, 8, 24, and 48 h after the infusion on Day 1
Volume of distribution at steady state (Vss) of FVIII | Samples taken prior and then 0.5, 4, 8, 24, and 48 h after the infusion on Day 1
Maximum Plasma Concentration (Cmax) of FVIII | Samples taken prior and then 0.5, 4, 8, 24, and 48 h after the infusion on Day 1
Minimum Plasma Concentration (Cmin) of FVIII | Samples taken prior and then 0.5, 4, 8, 24, and 48 h after the infusion on Day 1
Time the maximum concentration occurs (tmax) of FVIII | Samples taken prior and then 0.5, 4, 8, 24, and 48 h after the infusion on Day 1
Total clearance of the drug from the body (CL=dose/AUC) of FVIII | Samples taken prior and then 0.5, 4, 8, 24, and 48 h after the infusion on Day 1
Number of infusions per bleeding event | 1 day
Number of infusions per month | 1 month
Number of infusions per year | 1 year
Dose (IU/kg) per bleeding event | 1 day
Dose (IU/kg) per month | 1 month
Dose (IU/kg) per year | 1 year

SECONDARY OUTCOMES:
Frequency of adverse events (AEs) | 6 months
Severity of AEs per subject | 6 months
Severity of AEs per infusion | 6 months
Relatedness of AEs per subject | 6 months
Relatedness of AEs per infusion | 6 months
Development of FVIII inhibitors | Samples taken at screening visit, on day 2, on months 1 and 3, and at final visit

CONTACTS AND LOCATIONS:
Overall Officials: Program Director Clinical R&D, Study Director — CSL Behring
Locations (8):
- Belarus (2):
  - Study site, Homyel
  - Study site, Minsk
- Study Site, Tbilisi, Georgia
- Study Site, Guatemala City, Guatemala
- Study Site, Beirut, Lebanon
- Study site, Monterrey, Mexico
- Ukraine (2):
  - Study Site, Dnipropetrovsk
  - Study Site, Lviv